CLINICAL TRIAL: NCT03989869
Title: Very Early Medical Abortion - a Randomised Controlled Trial
Brief Title: Very Early Medical Abortion
Acronym: VEMASCOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Lothian (Other Government)
Collaborators: Karolinska Institutet (Other); University of Edinburgh (Other)
Responsible Party: Principal Investigator, John Reynolds-Wright, Clinical Research Fellow, University of Edinburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC19007; 257387 (Other: IRAS (NHS Ethics))
Record Dates: First submitted 2019-06-17; First posted 2019-06-18 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Abortion Early

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VEMA (Experimental): Immediate medical abortion treatment
  Interventions: Other: Immediate treatment
- Standard of Care (No Intervention): Delayed care until an intrauterine pregnancy has been confirmed with ultrasound.

INTERVENTIONS:
Other: Immediate treatment — Early Medical Abortion treatment, when ultrasound does not yet have conclusive signs of intrauterine pregnancy
  Arms: VEMA

SUMMARY:
The research question begin addressed by this study is "Is Very Early Medical Abortion (VEMA - before a pregnancy is visible on ultrasound scan) as effective as medical abortion when performed later and an intrauterine pregnancy can be visualised with ultrasound?".

This is important to patients and public, because delays to abortion care can cause mental distress, and pain and bleeding are worse at later gestations.

The study is examining whether earlier or delayed administration of abortion medications affects the efficacy and side effects of the medical abortion process, in women with very early pregnancies.

Any women who had a positive pregnancy test, requesting abortion, but did not have a visible pregnancy on ultrasound scan could take part in the study. Women with signs, symptoms or ultrasound findings suggesting ectopic pregnancy would not be included.

This study will be conducted at a community sexual and reproductive health centre that provides abortion care.

The participants will be involved in the study for a maximum period of 4 weeks. They will be randomly allocated to either immediate abortion care or delayed abortion care. In each arm of the study they will receive clinical care that they would otherwise routinely receive. In addition to this, they will receive a telephone call follow up with a short questionnaire to complete over the phone.

This study is being conducted in Scotland but the results will be combined with findings from similar research groups across Europe as part of a consortium of researchers. This consortium is coordinated by the Karolinska Institutet in Sweden under the EuDRACT ID: 2018-003675-35

ELIGIBILITY:
Inclusion Criteria:

1. Women 18 years old or above opting for medical abortion with a pregnancy estimated by gynaecological history and Last Menstrual Period (LMP - if known) to be less than 6 weeks
2. No signs of ectopic pregnancy, miscarriage or other pathological pregnancy
3. Transvaginal ultrasound (part of the clinical protocol at the abortion visit) shows no confirmed Intrauterine Pregnancy (IUP see definitions below)
4. Willing and able to return to the clinic for possible delayed treatment and at 1 to 2 weeks after the start of treatment for follow up
5. Capable of giving their informed consent to participate.

Exclusion Criteria:

1. Women with visible (confirmed) IUP
2. Women with contraindications to medical abortion including diagnosed pathological pregnancy at the initial examination.
3. Inability to give informed consent.

The following definitions will be used according to the consensus statement on nomenclature, definitions and outcomes in pregnancy of unknown location (Barnhart et al, Fertil Steril. 2011;95:857-66):

1. Confirmed IUP: Ultrasound shows an intrauterine yolk sac or fetal structure with or without cardiac echo.
2. Not confirmed IUP: This group includes cases where:

   1. ultrasound shows an empty uterine cavity (frequently referred to as PUL: Pregnancy of Unknown Location) or
   2. ultrasound shows a gestational sac, or sac like structure, but without a yolk sac.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Complete Abortion Rate (efficacy) | Within 30 days of treatment initiation
  Rate of complete abortion without surgical intervention, as reported by patients using a self-administered low-sensitivity pregnancy test at 2 weeks after treatment. This will be collected via telephone questionnaire.

SECONDARY OUTCOMES:
Complication Rate | Within 30 days of treatment initiation
  Rate of complications including ectopic pregnancy, infection.
Duration of post-abortion bleeding | Within 30 days of treatment initiation
  Number of days bleeding following treatment
Acceptability of method | Within 30 days of treatment initiation
  Preference for delay or immediate treatment
Visual Analogue Pain score | Within 30 days of treatment initiation
  Visual Analogue Scale of pain experienced during abortion. Mean will be reported and range of scale from 0-10.

CONTACTS AND LOCATIONS:
Overall Officials: John J Reynolds-Wright, MBChB, Principal Investigator — NHS Lothian and University of Edinburgh
Locations (1):
- Chalmers Centre for Sexual and Reproductive Health, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data will be shared with our collaborators at Karolinska Institutet but not publically available.

REFERENCES:
- [Derived] Gyllenberg F, Brandell K, Jar-Allah T, Kallner HK, Reynolds-Wright J, Boerma C, Cameron S, Hognert H, Heikinheimo O, Kaislasuo J, Gemzell-Danielsson K. Differences in pain, bleeding, and satisfaction during medical abortion at very early gestations. Acta Obstet Gynecol Scand. 2025 Sep;104(9):1665-1671. doi: 10.1111/aogs.15177. Epub 2025 Jul 2. PMID 40600383
- [Derived] Brandell K, Jar-Allah T, Reynolds-Wright J, Kopp Kallner H, Hognert H, Gyllenberg F, Kaislasuo J, Tamang A, Tuladhar H, Boerma C, Schimanski K, Gibson G, Lokeland M, Teleman P, Bixo M, Mandrup Kjaer M, Kallfa E, Bring J, Heikinheimo O, Cameron S, Gemzell-Danielsson K; VEMA (Very Early Medication Abortion) Study Group. Randomized Trial of Very Early Medication Abortion. N Engl J Med. 2024 Nov 7;391(18):1685-1695. doi: 10.1056/NEJMoa2401646. PMID 39504520